CLINICAL TRIAL: NCT06783413
Title: Effects of Laughter Yoga on Fatigue, Sleep Quality and Psychological Well-Being in Patients With Multiple Sclerosis: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Principal Investigator, Nurgül KAPLAN, Sponsor-Investigator, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GaziosmanpasaU- HMŞRLK-NK-02
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis; Fatigue; Sleep Quality; Psychological Well-being
Keywords: Multiple Sclerosis; Laughter Yoga; Fatigue; Sleep Quality; Psychological Well-Being; Nursing
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Sleep Initiation and Maintenance Disorders; Psychological Well-Being | interventions — Laughter Therapy; Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized-controlled
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know which group they are in. The person who analyzes the data obtained at the end of the study will not know
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group( Laughter Yoga Group) (Experimental): This group will participate in laughter yoga sessions twice a week for 30 minutes. These sessions include breathing techniques, laughter exercises and relaxation activities. The intervention period is 6 weeks in total.
  Interventions: Behavioral: Intervention group (Laughter Yoga)
- No Intervention (Control Group) (Other): Participants in the control group will undergo standard care procedures without receiving any intervention. The results will be evaluated for comparison purposes.
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Intervention group (Laughter Yoga) — Laughter yoga is a practice that includes physical laughing exercises and breathing techniques. Sessions will be conducted as group therapy with a trained guide. The intervention will be applied to evaluate changes in participants' fatigue, sleep quality and psychological well-being.
  Arms: Intervention Group( Laughter Yoga Group)
Other: Control group — Participants in the control group will continue to receive their current standard of care and will not receive any additional interventions.
  Arms: No Intervention (Control Group)

SUMMARY:
This study is planned to evaluate the effects of laughter yoga applied to patients with multiple sclerosis on fatigue, sleep quality and psychological well-being.

Although there are studies in the national and international literature that separately address the effects of laughter therapy on fatigue, sleep quality and psychological well-being, no studies have been found that address the effects of laughter therapy on fatigue, sleep quality and psychological well-being in patients with multiple sclerosis. This study is expected to make a significant contribution to the literature as it is the first experimental study to evaluate the effects of laughter therapy and laughter yoga applied to patients with multiple sclerosis on fatigue, sleep quality and psychological well-being. It is also thought that this study can guide studies to be conducted with other parameters. This study is planned to evaluate the effects of laughter yoga applied to patients with multiple sclerosis on fatigue, sleep quality and psychological well-being.

Research Hypothesis H1: Laughter yoga reduces the fatigue level of multiple sclerosis patients compared to the control group.

H2: Laughter yoga increases the sleep quality of multiple sclerosis patients compared to the control group.

H3: Laughter yoga increases the effect of laughter yoga on psychological well-being of multiple sclerosis patients compared to the control group.

Variables of the Study Dependent Variables: Introductory Information Form, Fatigue Severity Scale-YSQ, Pittsburgh Sleep Quality Index (PSQI), Psychological Well-Being Scale (PWSS) and Expanded Disability Status Scale (EDSS) will be used.

Independent Variables: Laughter Yoga

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a neurological disease characterized by inflammation and demyelination in the central nervous system and is seen in young adults (Yeni et al., 2022). MS usually begins between the ages of 20-40, and is three times more common in women than in men (Ford, 2020). According to the 2020 data of the Multiple Sclerosis International Federation (MSIF), it has been reported that MS has reached 2.8 million people worldwide (MSIF, 2020). In MS, many symptoms are observed due to the deterioration of nerve conduction due to myelin sheath and axon damage; as the disease progresses, the symptoms cause permanent damage and restrictions in the individual's physical, emotional and social life (Yeni et al., 2022). In MS, 70-80% of patients have MS-related fatigue, and more than 55% report that the worst symptom is fatigue. When fatigue is seen together with other symptoms, it causes an increase in disability, deterioration in quality of life and negatively affects daily life activities (Miller & Soundy, 2017). The etiology of fatigue, which can also be defined as physical or mental energy deficiency and weakness in the literature, is not fully known; multifactorial etiology with individual, environmental and developmental causes is mentioned (Hür & Sezgin, 2017; Pekçetin et al., 2019). Fatigue is a subjective finding and many factors (neurological dysfunctions, anxiety, depression, pain, spasticity, sleep disorders, medications, etc.) are involved in its physiopathology. Nonpharmacological methods provide great benefits in coping with fatigue. It has been reported that the most studied nonpharmacological method in coping with fatigue in MS patients is physical exercise (Yeni et al., 2022). Sleep disorders are quite common in people with MS due to fatigue, pain and deterioration in quality of life. Sleep is considered a critical brain condition for motor learning and memory consolidation, and there is a need for practices to improve sleep quality in individuals with MS (Al-Sharman et al., 2019). The concept of psychological well-being has been defined as "managing existential challenges faced in life (such as pursuing meaningful goals, personal development, and establishing quality relationships with others)" (Keyes et al., 2002). Multiple sclerosis affects the central nervous system, causing many psychological problems that affect patients' psychological health as well as physical problems (Malekzadeh et al., 2020). According to the World Health Organization (WHO); "traditional medicine has a long history. Laughter, which is a natural part of our lives, is a natural, sincere, innate, universal response that we give as a response to humorous stimuli. Laughter and yoga are combined with breathing techniques and are used in the field of complementary medicine today as "Laughter Yoga" (Öztürk and Tezel, 2021). In addition to medical treatment, traditional and complementary medicine (GETAT) methods and sleep quality disorders are used in the treatment (Turan et al., 2010). Laughter Yoga, one of the types of yoga, was developed by Indian physician Dr. Madan Kataria in 1995 and each session consists of breathing exercises, stretching-relaxation techniques and laughter exercises (Yazdani et al., 2014). Laughter yoga, which can be applied by nurses as a noninvasive method, is a complementary and alternative treatment method that aims to develop and improve the health of individuals (Karali E, 2020). Laughter yoga, which is a very innovative application, is used in nursing to reduce anxiety, stress and fatigue levels, reduce pain, improve mental functions, and increase sleep and quality of life (Öztürk, 2018). Studies have reported that laughter yoga is usually applied once or twice a week, with sessions of 30-45 minutes; 4, 8 and 12 sessions (Kin et al., 2017). Laughter yoga can only be practiced by people who have received a "Laughter Yoga" certificate, and the role of the practitioner is very important (Kuru, 2016). Laughter causes effects such as a decrease in blood pressure and muscle tension, an increase in saturation value, respiratory rate and happiness hormones, a decrease in stress hormones, and an improvement in the immune system and mental processes in our bodies (Yım, 2016). Laughter yoga is recommended for hemodialysis patients to reduce pain, anxiety, depression and fatigue; and to increase immunity, quality of life and sleep quality (Bennett et.al., 2014). According to the results of the study, it has been proven that it has positive effects in terms of body and soul and it is thought that it can be used in different areas of health.

Data Collection Tools The research will use the following data collection tools: Introductory Information Form, Fatigue Severity Scale-YSÖ, Pittsburgh Sleep Quality Index (PSQI), Psychological Well-Being Scale (PSS) and Expanded Disability Status Scale-EDSS.

Introductory Information Form The 'Introductory Information Form' developed by the researcher includes questions regarding the participants' age, marital status, education level, employment status, type of multiple sclerosis, number of years of multiple sclerosis, presence of a disease other than multiple sclerosis, having had a multiple sclerosis attack in the last 6 months, having undergone surgery in the last 6 months, and presence of a psychiatric diagnosis.

Fatigue Severity Scale-YSÖ The validity and reliability of the scale developed by Krupp et al. (1989) was tested in 2007 by Armutlu et al. (Krupp et al., Armutlu et al., 2007). It is a 7-point Likert-type scale consisting of nine items. Each item is defined as 1 = completely disagree, 7 = completely agree. The lowest score possible from the scale is 9 and the highest is 63, and as the scale score increases, the level of fatigue also increases. The Cronbach alpha value of the scale was found to be 0.94 (Armutlu et al., 2007).

Pittsburgh Sleep Quality Index (PSQI) The Pittsburgh Sleep Quality Index (PSQI) was created by Buyyse et al. in 1989. Its validity and reliability studies in Turkey were conducted by Ağargün et al. in 1996. The PSQI consists of a 24-question survey that evaluates sleep quality and disorders by scoring them over a one-month period. 19 of the questions are answered individually, and 5 questions are answered by the individual's family or a roommate. The questions in the survey are divided into 7 components. Each component is evaluated between 0-3 points. An increase in the PSQI score and a total PSQI score of 5 and above indicates that sleep quality has deteriorated. The Cronbach alpha value of the PSQI was determined as 0.80 (Ağargün et al., 1996).

Psychological Well-Being Scale (PSWS) The scale was developed by Diener et al. (2010) to define important components of human functioning such as positive relationships, feelings of competence, and the ability to live a meaningful and purposeful life, and consists of eight items (Diener et al., 2010). The Turkish adaptation of the scale was made by Telef (2013). The scale is a 7-point Likert-type scale ranging from strongly disagree (1) to strongly agree (7). All items are expressed positively. The lowest score is 8, and the highest score is 56. A high score indicates that the individual has many psychological resources and strengths. In the reliability study conducted by Telef, Cronbach's Alpha value was determined as 0.80 (Telef, 2013).

Expanded Disability Status Scale (EDSS) It was developed by Kurtzke (1983) to evaluate disability status. Pyramidal, cerebellar, brainstem, sensory, visual, bowel-bladder functions and mental functions are evaluated and the EDSS score is calculated. The rating is made according to the best performance the patient can show without excessive effort, and 0-4 points indicate that the patient is independent, 6.0 points indicate unilateral support and 7.0 points and above indicate dependence on a wheelchair or bed. Patients score between 0-10 on this scale and the degree of disability increases as the score increases (Kurtzke, 1983).

Data Collection Patients between the ages of 18-65 who are diagnosed with MS according to McDonald criteria and are followed up by the MS outpatient clinic of the Neurology Department of Tokat Gaziosmanpaşa University Hospital will be referred to the researcher by their neurology specialist physician. Patient interviews are planned to be conducted in the outpatient clinic. Patients who are referred to the researcher by the physician and who agree to participate in the study and who meet the sample selection criteria will be randomized and included in the study by determining the control and intervention groups. It is planned to apply data collection tools to all patients who agree to participate in the study (control and intervention groups) after the purpose of the study is explained during the first interview and verbal and written consent is obtained.

Pre-test data: It was planned to collect pre-test data by informing the patients who meet the inclusion criteria. In the study, the Introductory Information Form, Fatigue Severity Scale-YSQ, Pittsburgh Sleep Quality Index (PSQI) and Psychological Well-Being Scale (PWS) will be used as data collection tools. It was planned to inform the patients that they would be asked to fill out the questionnaires again at the end of 6 weeks.

Post-test data: 6 weeks after the pre-test data is collected, the link will be shared with the patients online via WhatsApp to apply the measurement tools to be used in collecting the post-test data, and they will be asked to fill out the forms. Fatigue Severity Scale-YŞÖ, Pittsburgh Sleep Quality Index (PSQI), Psychological Well-Being Scale (PWW) will be included in the link.

In this study, it is planned to apply laughter yoga to the patients in the intervention group twice a week for six weeks, for a total of 12 sessions. Laughter yoga sessions will be held via the Zoom program. A WhatsApp group will be established to facilitate communication with the patients before starting laughter yoga, and information about the sessions will be shared via the group. It is planned for the patients in the intervention group to download the Zoom program before the application. Since the more participants there are in laughter yoga, the more laughter spreads and the easier it will be for the participants to laugh, it is recommended that laughter yoga sessions be held in groups and that each group consists of at least five people to ensure group dynamics. It is planned to create groups by determining appropriate time intervals for patients to participate online. It is planned to contact patients via phone to avoid disruptions in the sessions. No intervention will be made to patients in the control group during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Being between the ages of 18-65
2. Being literate
3. Being diagnosed with MS
4. Not having had an attack in the last month
5. Being under 6.5 on the Expanded Disability Status Scale (EDSS)
6. Not having a diagnosis of cognitive or mental disorder
7. Being willing to participate in the study
8. The patient has internet access
9. Not having incontinence

Exclusion Criteria:

1. Having a diagnosis of cognitive or mental disorder
2. Having communication problems
3. Having previously experienced laughter yoga
4. Having a history of surgery in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Fatigue | 6 weeks
  Change in fatigue levels measured using the Fatigue Severity Scale (FSS). Participants' fatigue scores will be assessed at baseline and at the end of 6 weeks to assess the effectiveness of laughter yoga.

SECONDARY OUTCOMES:
Sleep Quality | 6 weeks
  Change in sleep quality measured using the Pittsburgh Sleep Quality Index (PSQI). Sleep scores will be assessed at baseline and at the end of 6 weeks to assess the effect of laughter yoga.

OTHER OUTCOMES:
Effect on Psychological Well-Being | 6 weeks
  Assessment of changes in psychological well-being using the Psychological Well-being Scale (PWBS). The assessment will focus on areas such as self-acceptance, positive relationships, autonomy, environmental mastery, purpose in life, and personal growth. Scores will be compared at baseline and Week 6 to determine the impact of the intervention on psychological well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR